CLINICAL TRIAL: NCT02055560
Title: Retrospective Data Comparison of Toxicity and Efficacy in Colorectal Cancer (CRC) Patients Managed With and Without 5-FU Exposure Optimization Testing
Brief Title: Retrospective Evaluation of 5-FU Exposure Optimization in CRC Patients
Acronym: 5-FU RECORD
Status: Completed | Type: Observational
Sponsor: Saladax Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SBI-5FU-005
Record Dates: First submitted 2014-01-31; First posted 2014-02-05 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Metastatic Colorectal Cancer; Adjuvant Colorectal Cancer; 5-FU Containing Therapy Regimens
Keywords: colorectal; OnDose; MyCare; 5-FU; pharmacokinetics; exposure; optimization; dose adjustment
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PK-Guided Cohort: CRC patients who were treated with 5-FU containing therapy regimen where 5-FU dosing was monitored and optimized using PK-guided dose adjustment.
- BSA Cohort: CRC patients who were treated with 5-FU containing therapy regimen where 5-FU dosing was done according to body surface area (BSA) and no PK monitoring was performed.

SUMMARY:
The primary objective of this study is to evaluate whether the management of colorectal cancer (CRC) patients with 5-fluorouracil (5-FU) exposure optimization testing reduces 5-FU related toxicities and improves outcomes compared to the current standard of care. A secondary objective is to characterize the variability of 5-FU levels among CRC patients managed with 5-FU exposure optimization testing and the impact of such management on 5-FU plasma levels and drug doses during the course of chemotherapy.

DETAILED DESCRIPTION:
This is a multi-center retrospective matched cohort study of early and late stage CRC patients who received 5-FU doses determined using body surface area (BSA) and in patients who underwent pharmacokinetically (PK)-guided 5-FU dose monitoring and adjustment. A retrospective chart / electronic medical record review of colorectal cancer patients treated with infusional 5-FU regimens between May 1, 2009 and December 31, 2013, satisfying the inclusion/exclusion criteria, will be performed. In this multi-center study, patients who underwent PK-testing during at least two different 5-FU administrations will be matched to patients who received doses based on their BSA, treated at the same institution. Matching for selection of the BSA cohort at each site will be done using the following criteria (based on factors that may influence 5-FU metabolism): age, gender, disease stage, prior chemotherapy treatment, and 5-FU containing treatment regimen being used. Each patient will be assigned a random five-digit Study ID number to protect patient confidentiality. Minimal medical history/demographics data will be collected from the patient's medical records / clinic chart using paper case report forms (CRFs). The data to be collected from each patient's records will include: patient demographics (i.e. gender, age, height, and race), colorectal cancer diagnosis (i.e. date of primary diagnosis, tumor stage, grade, histology and phenotype, and date of metastatic diagnosis and sites of metastases if applicable), use of prior therapies for treatment of CRC, 5-FU containing regimen details throughout the 5-FU treatment (i.e. weight, BSA, ECOG status, doses of each drug used in the regimen, and 5-FU infusion start/stop dates and times), 5-FU PK testing results (if applicable), concomitant procedures and medications, CBC and chemistry testing results, adverse events experienced during 5-FU therapy regimen, and tumor response and follow-up information. Patients will not be contacted for the purposes of this study and a waiver of HIPAA authorization will be requested from the appropriate IRB. Once data has been collected and monitored, all records tying the random Study ID number to a specific patient at the sites will be destroyed, rendering all information de-identified.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years of age or older.
* Patients with histologically confirmed colorectal cancer who were treated with an infusional 5-FU regimen between May 1, 2009 and December 31, 2013.
* PK-Guided Cohort: Patients monitored with 5-FU PK-testing at a minimum of two administrations of 5-FU throughout the course of a single infusional 5-FU containing treatment regimen.
* BSA Cohort: Patients who received infusional 5-FU doses calculated based on their BSA.

Exclusion Criteria:

* Patients less than 18 years of age.
* Patients with concurrent treatment of other active malignancies.
* Patients that underwent radiation therapy concurrently with chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients treated with 5-FU containing therapy regimens by US based oncologists in community and academic setting. Sites which ordered >20 Myriad OnDose tests in 2012 will be approached for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-04-02 (Actual); Study Completion 2015-12-18 (Actual)

PRIMARY OUTCOMES:
Variability of 5-FU plasma levels (exposure) | At each cycle after initiation of 5-FU containing therapy, or approximately every 1 - 2 weeks, depending on the 5-FU infusion schedule, for up to ~12 cycles (~24 weeks) total.
  At each treatment cycle (i.e. Cycle 1, Cycle 2, Cycle 3, etc.), we will plot the 5-FU exposure (i.e. AUC value) and determine the average, median, standard deviation, and percent coefficient of variation (%CV). These statistics will also be determined for all 5-FU exposure values combined.
Hematological and non-hematological toxicity rates | From initiation of the 5-FU containing therapy until up to 30 days after its discontinuation, or for up to ~28 weeks total
  Incidence of 5-FU related toxicities, such as diarrhea, oral mucositis, neutropenia, anemia, febrile neutropenia, thrombocytopenia, nausea, etc., will be recorded throughout the duration of the 5-FU containing therapy regimen.
Tumor response | At each follow-up disease assessment following initiation of 5-FU containing thearpy, expected to occur an average of every 8 - 12 weeks, until discontinuation of therapy, or up to ~24 weeks total.
  Tumor response rates as determined by imaging [classified as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD)].
Progression-free survival (PFS) | up to 3.5 years after initiation of 5-FU containing therapy regimen
Overall survival | up to 3.5 years after initiation of 5-FU containing therapy regimen

CONTACTS AND LOCATIONS:
Overall Officials: Craig Miller, B.S., Study Director — Saladax Biomedical, Inc.
Locations (5):
- United States (5):
  - University of California San Diego, La Jolla, California
  - Hematology/Oncology of the North Shore, Skokie, Illinois
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Tennessee Plateau Oncology, Crossville, Tennessee
  - Texas Health Physicians Group, Plano, Texas

IPD SHARING:
Plan to Share IPD: No